CLINICAL TRIAL: NCT06483997
Title: Associations Between Diet, Hepcidin, and Relative Dose Intensity Among Women Receiving Chemotherapy for Breast or Gynecological Cancer
Brief Title: Diet, Hepcidin, and Chemotherapy RDI
Status: Active, not recruiting | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Kimberly Robien, Associate Professor, George Washington University
Other Study IDs: NCR245680
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Female; Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Endometrial Cancer; Gynecologic Cancer
Keywords: nutrition; inflammation; anemia; toxicity; chemotoxicity
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Inflammation; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, observational cohort study will evaluate the extent of associations between self-reported pro- or anti- inflammatory dietary intake patterns for one month before induction chemotherapy for gynecological cancer or neo/adjuvant chemotherapy for breast cancer and baseline serum hepcidin concentrations. Associations between hepcidin concentration and relative dose intensity (RDI) of chemotherapy will also be evaluated.

DETAILED DESCRIPTION:
This is a prospective, observational cohort of 100 women receiving chemotherapy for breast or gynecological cancer at GW Cancer Center from July 1, 2024 - approximately September 2025. At study baseline (after diagnosis, but prior to starting chemotherapy), participants will complete a ~30-minute food frequency questionnaire (FFQ) and demographic/food security survey using a preprogrammed iPad in the clinic. The clinical research nurse will obtain an additional research blood draw at the same time as the patient's routine clinical blood draw prior to chemotherapy initiation for serum hepcidin concentration measurement. Data on cancer type, premorbid medical conditions, and chemotherapy plans and administration will be collected from the electronic health record by study staff and the duration of data collection will be the length of chemotherapy plus 30 days. Data will be used to address the objectives below.

Among adult women scheduled to receive chemotherapy for breast or gynecological cancer treatment, the objectives/aims of this study will be to:

1. Determine the extent to which pretreatment, self-reported Dietary Inflammatory Index dietary pattern scores from dietary intake during the one month prior to chemotherapy initiation are associated with pretreatment serum hepcidin concentrations
2. Determine the extent to which pretreatment serum hepcidin concentrations are associated with chemotherapy RDI.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with invasive breast cancer, OR
* Have been diagnosed with epithelial ovarian cancer, fallopian tube or primary peritoneal cancer, OR
* Have been diagnosed with endometrial cancer
* Are chemotherapy-naïve
* Are scheduled to receive neoadjuvant chemotherapy (or adjuvant chemotherapy following lumpectomy for breast cancer patients) or neoadjuvant/induction chemotherapy for gynecological cancer at GW Cancer Center

Exclusion Criteria:

* Prior primary hematological condition that would cause abnormal blood counts (e.g. leukemia)
* Pregnant at the time of potential enrollment
* Receipt of erythropoietin-stimulating agents or blood transfusion in the 6 weeks prior to initial testing
* Women who are cognitively unable to provide a diet history for the month prior to assessment.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 women receiving chemotherapy for breast or gynecological cancer at GW Cancer Center from July, 2024 - July, 2026
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Serum hepcidin concentration | pre-chemotherapy, single measure
  ng/ml, continuous
Chemotherapy relative dose intensity | during chemotherapy (up to 6 months, depends on duration of chemotherapy regimen), represents repeated measures
  Calculated variable that represents the ratio of chemotherapy actually received during the duration of treatment to the planned chemotherapy dose during the planned duration

SECONDARY OUTCOMES:
Hematologic toxicity | at any point during chemotherapy or within 30 days after completion of chemotherapy (up to 6 months, depends on length of chemotherapy regimen)
  Incidence of CTCAE grade 3 or higher hematologic toxicity (anemia, neutropenia, thrombocytopenia)
Treatment delays | at any point during chemotherapy (up to 6 months, depends on length of chemotherapy regimen)
  Delay of chemotherapy due to chemo-related adverse events, including hematologic toxicity, infection, hospitalization, or severe symptoms
Treatment change or discontinuation | at any point during chemotherapy (up to 6 months, depends on length of chemotherapy regimen)
  Change of chemotherapy regimen or discontinuation of treatment due to chemo-related adverse events, including hematologic toxicity, infection, hospitalization, or severe symptoms
Blood transfusion | at any point during chemotherapy or up to 30 days after completion of chemotherapy (up to 6 months, depends on length of chemotherapy regimen)
  Infusion of red blood cells, platelets, fresh frozen plasma, or other donated human blood products due to chemo-related hematologic toxicity
Hospitalizations | at any point during chemotherapy or up to 30 days after completion of chemotherapy (up to 6 months, depends on length of chemotherapy regimen)
  Unscheduled admission to a hospital or similar medical facility due to due to chemo-related adverse events, including hematologic toxicity, infection, or severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kim Robien, PhD, RD, Principal Investigator — Milken Institute School of Public Health, George Washington University
Locations (1):
- George Washington University Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may contact the PI with proposals to collaborate on secondary analyses using the study data. To protect participants privacy and data security, no individual patient data will be made available to external researchers.

DOCUMENTS (1):
  • Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT06483997/ICF_000.pdf